CLINICAL TRIAL: NCT06898944
Title: Analysis for Prognosis and Risk Factors for Acute Kidney Injury: Multi-center Cohort Study
Brief Title: Prognosis and Risk Factors for Acute Kidney Injury
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); SMG-SNU Boramae Medical Center (Other); Keimyung University Dongsan Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: H-2208-015-1347
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- AKI group: * Aged 20 years or older who visited hospital
  * Underwent at least two blood tests, including serum creatinine, within an interval of 7 days or less
  * AKI was defined based on the KDIGO criteria (an increase in serum creatinine by ≥0.3 mg/dL or ≥1.5 times the baseline).
- Control group: Control group was matched 1:1 to the AKI group based on age, sex, year of visit, and baseline kidney function, forming the study population.

SUMMARY:
The aim of our study is to analyze the accurate diagnosis and prognosis of acute kidney injury (AKI) based on its severity and to define long-term clinical and socioeconomic outcomes.

Investigators defined the AKI group among adults aged 20 years or older who visited enrolled center and underwent at least two blood tests, including serum creatinine, within an interval of 7 days or less and a control group was matched 1:1 to the AKI group based on age, sex, year of visit, and baseline kidney function, forming the study population. Investigators then collected and analyzed various clinical, laboratory, and hospitalization records including demographic data, anthropometric data, laboratory data, and medical history.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 20 years old who visited Parcitipating Medical Center (Seoul National University Hospital, Bundang Seoul National University Hospital, SMG-SNU Boramae Medical Center, Keimyung University Dongsan Medical Center) between 2006 and 2021
* The AKI group is defined as individuals meeting the AKI diagnostic criteria of the KDIGO Guideline (an increase in serum creatinine of ≥0.3 mg/dL or ≥1.5 times the baseline level) is enrolled.
* The Control Group is defined as individuals from the study population who do not meet the AKI criteria and are matched 1:1 based on age, sex, year of visit, and baseline renal function.

Exclusion Criteria:

* Individuals under 20 years old
* Individuals who did not undergo serum creatinine tests meeting the criteria
* Individuals with pre-existing end-stage kidney disease (ESKD) who have undergone dialysis or kidney transplantation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥20 years old) who visited Parcitipating Medical Center (Seoul National University Hospital, Bundang Seoul National University Hospital, SMG-SNU Boramae Medical Center, Keimyung University Dongsan Medical Center) between 2006 and 2021
Sampling Method: Non-Probability Sample
Enrollment: 320000 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Serum Creatinine | From Index Date(The Date Which Acute Kidney Injury Occured) Through 5 Years After The Index Date

SECONDARY OUTCOMES:
Change from Baseline in Urine Protein/Creatinine Ratio | From Index Date(The Date Which Acute Kidney Injury Occured) Through 5 Years After The Index Date
Incidence of Receiving Renal Replacement Therapy | From Index Date(The Date Which Acute Kidney Injury Occured) Through 5 Years After The Index Date
Change from Baseline in Serum Hemogloblin Level | From Index Date(The Date Which Acute Kidney Injury Occured) Through 5 Years After The Index Date
Change from Baseline in Serum Albumin Level | From Index Date(The Date Which Acute Kidney Injury Occured) Through 5 Years After The Index Date

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ki Kim, M.D. Ph.D., Principal Investigator — Department of Internal Medicine, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes